CLINICAL TRIAL: NCT05254964
Title: Effect of Intensive Cognitive Rehabilitation on Cognitive, Motor, and Language Functional Networks in Subacute Stroke Patient
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients not recruited.
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12-019
Record Dates: First submitted 2022-02-09; First posted 2022-02-24 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Cognitive Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive cognitive rehabilitation group (Experimental): Participants receive intensive cognitive rehabilitation for 20 hours for 4 weeks.
  Interventions: Procedure: Cognitive rehabilitation

INTERVENTIONS:
Procedure: Cognitive rehabilitation — Intensive cognitive rehabilitation by cognitive therapist for 1 hour on every working 20 days (4 weeks) during the subacute stroke phase

SUMMARY:
Altered brain networks, including cognitive, motor, and language networks, are investigated by intensive cognitive rehabilitation in subacute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 to 80 years
* Patients with subacute stroke within 2 weeks of onset
* First-ever stroke
* Supratentorial stroke
* Less than 8 SAFE (shoulder abduction, finger extension) points
* Less than 35 FMA Upper scores
* MEP (motor evoked potential) negative
* Not more than 24 K-MMSE (Korean Mini-Mental State Examination) score

Exclusion Criteria:

* Difficult to communicate due to severe language impairment.
* Accompanied by an existing serious neurogenic disease
* Existing significant psychiatric disorders such as major schizophrenia, bipolar disorder
* If there are difficulties in conducting the research
* Any patients who are judged by the investigator to be difficult to participate in this study
* Patients with contraindicated MRI scans

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Strength of connectivity in brain network obtained from MRI neuroimaging data | Change in strength of connectivity after intensive cognitive rehabilitation for 4 weeks
  Participants' MRI neuroimaging data are acquired at pre- and post-intervention. Brain network can be constructed using MRI neuroimaging data, and strength of connectivity can be calculated in the brain network. Strength of connectivity has a value between -1 and 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea